CLINICAL TRIAL: NCT01935128
Title: A 24-month, Single Center, Pilot, Open Label, Controlled Trial to Evaluate the Efficacy and Safety of Calcineurin-inhibitor Reduction With Conversion at 2 Months to Reduced Dose Tacrolimus/Everolimus in Adult Renal Transplant Recipients Following Campath® Induction and Steroid Avoidance
Brief Title: Evaluation of Calcineurin-inhibitor Reduction With Conversion at 2 Months to Everolimus/Reduced Tacrolimus in Renal Transplant Recipients Following Campath® Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michael A. Rees, MD, PhD, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Everolimus
Record Dates: First submitted 2013-08-21; First posted 2013-09-04 (Estimated); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Renal Transplant
Keywords: Renal Transplant; Immunosuppression; Steroid Avoidance; Calcineurin Avoidance; Mammalian Target of Rapamycin (mTOR); Kidney
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 Everolimus/Reduced dose tacrolimus (Experimental): In this arm, the myfortic® will be weaned off quickly and everolimus (Zortress®) initiated to achieve a target level of 3-8 ng/ml with a mean of 6 ng/ml. Once achieving a therapeutic dose of everolimus (Zortress®) the tacrolimus (Prograf® or Hecoria®) dose will be reduced a target level of 3-5 ng/ml.
  Interventions: Drug: Arm 1 Everolimus/Reduced dose tacrolimus

INTERVENTIONS:
Drug: Arm 1 Everolimus/Reduced dose tacrolimus — Immunosuppression drug intervention
  Other Names: Zortress®; Prograf® or Hecoria®

SUMMARY:
The purpose of this study is to evaluate whether conversion to everolimus (Zortress®), allowing the elimination or reduction of calcineurin inhibitors, will reduce nephrotoxicity (measured by increased creatinine clearance) and lengthen overall graft (kidney transplant) survival (measured by 2-3 year graft survival).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether conversion to everolimus (Zortress®), allowing the elimination or reduction of calcineurin inhibitors, will reduce nephrotoxicity (measured by increased creatinine clearance) and lengthen overall graft (kidney transplant) survival (measured by 2-3 year graft survival). Among the worst of the long-term effects of chronic immunosuppression are the nephrotoxicity (toxic to kidney cells) of the calcineurin inhibitors and the myriad complications of steroids. This protocol evaluates the elimination or reduction of calcineurin inhibitors in a protocol that has already successfully eliminated the long-term use of steroids. A considerable need remains for safer therapeutic agents that inhibit T-cell activation (a white blood cell that attacks foreign cells as part of the immune response) via a calcineurin independent or reduced-dose mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Male or female renal allograft recipients at least 18 years old.
* Patients who have given written informed consent to participate in the study. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
* Patient who has received a kidney transplant from a deceased or living unrelated-/related donor.
* Recipient of a kidney allograft with a cold ischemia time (CIT) < 36 hours.
* Female patients must have a negative pregnancy test prior to study enrollment.
* Patients on calcineurin inhibitor(s) (CNI) (tacrolimus and myfortic®) without steroid maintenance following Campath® induction.
* Patients with an acceptable allograft function defined by a serum creatinine < 2.5 mg/dL (250 μmol/L) and an actual estimated glomerular filtration rate (eGFR) (Modification of diet in renal disease equation 4, MDRD4) ≥ 30 mL/min/1.73m2 (without renal replacement therapy).
* No evidence of rejection since the time of transplantation.

Exclusion Criteria:

* Recipient of ABO incompatible allograft or a positive cross-match.
* Patient who is human immunodeficiency virus (HIV) positive.
* Patient who received an allograft from a Hepatitis B surface Antigen (HBsAg) or a Hepatitis C Virus (HCV) positive donor.
* HBsAg and/or a HCV positive patient with evidence of elevated liver function tests (LFTs) (Alanine transaminase/Aspartate transaminase [ALT/AST] levels ≥ 2.5 times upper limit of normal [ULN]). Viral serology results obtained within 6 months prior to randomization are acceptable.
* Patient with severe restrictive (total lung capacity [TLC] < 50%) or obstructive pulmonary (forced expiratory volume in one second [FEV1] < 50) disorders.
* Patient with severe allergy requiring acute (within 4 weeks of baseline) or chronic treatment that would prevent patient from potential exposure to everolimus, or with hypersensitivity to drugs similar to everolimus (e.g. macrolides).
* Patients with a known hypersensitivity/contraindication to any of the immunosuppressants or their classes, or to any of the excipients.
* Patient with severe hypercholesterolemia (> 300 mg/dL) or hypertriglyceridemia (> 400 mg/dL) that cannot be controlled despite lipid lowering therapy.
* Patient with white blood cell (WBC) count ≤ 1,000 /mm3 (and absolute neutrophil count [ANC] of <500) or a platelet count ≤ 50,000 /mm3.
* History of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases. (Localized basal cell carcinoma of the skin at any time, or small (less than 4 cm) or low-grade renal cancers, bladder cancers, or treated prostate cancer with no evidence of disease after 2 years are allowable)
* Graft loss.
* Patient on renal replacement therapy.
* Patient who experienced biopsy proven rejection.
* Proteinuria > 1 g/day (as calculated from the urinary protein-to-creatinine ratio).
* Patients with recurrence of Focal Segmental Glomerulosclerosis (FSGS).
* Patient who has a current severe systemic infection according to the investigator judgment requiring continued therapy that would interfere with the objectives of the study.
* Patients with ongoing wound healing problems, clinically significant infection requiring continued therapy or other severe surgical complication in the opinion of the investigator.
* Presence of intractable immunosuppressant complications or side effects.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum human chorionic gonadotrophin laboratory test (>5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rees, MD, PhD, Principal Investigator — University of Toledo, HSC
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited following renal transplantation at a single transplant center. Participants were recruited between 2 and 6 months post-transplant. Date of first enrollment was July 3, 2013 and date of last enrollment was July 6, 2018.
Pre-assignment Details: 50 participants met the inclusion/exclusion criteria and were enrolled in the treatment arm.
Period: Overall Study
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Started | 50
Completed | 43
Not Completed | 7
Not completed — Death | 1
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.74 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Renal Function
Description: Renal function in patients will be assessed using glomerular filtration rate (GFR) as measured by the Modified Diet Renal Disease (MDRD) estimation.
  Glomerular filtration is the process by which the kidneys filter the blood, removing excess wastes and fluids. Glomerular filtration rate (GFR) is a calculation that determines how well the blood is filtered by the kidneys, which is one way to measure remaining kidney function. GFR is also used to find the stage of chronic kidney disease. Glomerular filtration rate is usually calculated using a mathematical formula that compares a person's size, age, sex, and race to serum creatinine levels. The higher the GFR number, the better the kidney function; the lower the GFR number, the worse the kidney function. A GFR of 60 or higher is in the normal range. A GFR below 60 may mean kidney disease. A GFR of 15 or lower may mean kidney failure.
Time Frame: 2 years
Population: Intent to treat population (all participants assigned to treatment arm). Last observation carried forward (LOCF) imputation method
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
mL/min/1.73 m2 | 65.70 (20.04)

2. Primary Outcome: Graft Survival
Description: Graft survival is defined as the percentage of kidney transplants still functioning at 2 years post baseline visit . One patient died of natural causes at 12 months with a functioning graft.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 49

3. Primary Outcome: Biopsy Proven Acute Rejection
Description: The percentage of patients with a treated biopsy-proven acute rejection (a co-primary endpoint) within the 2 year study time period
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 1

4. Primary Outcome: Patient Survival
Description: Patient survival is defined as the percentage of patients still surviving at 2 years post baseline visit
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 49

5. Secondary Outcome: Impaired Glucose Tolerance
Description: The number of patients with impaired glucose tolerance as indicated by fasting blood glucose levels, Hemoglobin A1C (HgbA1C) levels and the need for hypoglycemic medications
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 14

6. Secondary Outcome: Proteinuria
Description: The number of patients with proteinuria as defined by spot urine protein to creatinine ratio greater than 1.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 7

7. Secondary Outcome: Lipid Levels
Description: The number of patients with hyperlipidemia as defined by the development of new onset hyperlipidemia in the baseline negative patients and the number of baseline positive patients who required starting a new lipid-lowering medication or an increase in dose of their lipid-lowering medication over the course of the study
Time Frame: 2 years
Population: The overall number of participants analyzed was 50. This population was split into participants who were negative for hyperlipidemia at baseline and developed new onset hyperlipidemia (10) identified in Row 1 and participants who were baseline positive for hyperlipidemia but who required a new lipid-lowering medication or an increase in the dose of their lipid-lowering medication over the course of the study (40) as identified in Row 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants
  Baseline negative patients with new onset hyperlipidemia: number analyzed (Participants) | 10
  Baseline negative patients with new onset hyperlipidemia | 7
  Baseline positive patients started on new lipid-lowering medication or needing increase in dose: number analyzed (Participants) | 40
  Baseline positive patients started on new lipid-lowering medication or needing increase in dose | 19

8. Secondary Outcome: Mouth Ulcers
Description: The number of patients with stomatitis/aphthous ulcer
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 14

9. Secondary Outcome: Gastrointestinal Complaints
Description: The number of patients with gastrointestinal complaints as indicated by abdominal pain, nausea, vomiting or diarrhea not accounted for by a specific episode of illness such as gastroenteritis
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 22

10. Secondary Outcome: Leukopenia
Description: The number of patients with leukopenia as indicated by white blood cell count less than 1.0, absolute neutrophil count less than 500 or the need for exogenous granulocyte stimulating factor administration
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 1

11. Secondary Outcome: Thrombocytopenia
Description: The number of patients with thrombocytopenia as defined by platelet count less than 50
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 0

12. Secondary Outcome: Neurotoxicity
Description: The number of patients with neurotoxicity as evidenced by incidence of new onset seizure activity or tremors
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 1

13. Secondary Outcome: Pneumonitis
Description: The number of patients with pneumonitis as demonstrated by lung inflammation symptoms such as shortness of breath and/or cough requiring clinical intervention and management
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 3

14. Secondary Outcome: Cytomegalovirus
Description: The number of patients with Incidence of cytomegalovirus infection as defined by need for hospitalization
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 0

15. Secondary Outcome: Infection Requiring Hospitalization
Description: The number of patients with serious infections as defined by need for hospitalization
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 11

16. Secondary Outcome: BK Infection
Description: The number of patients with BK infection as defined by blood titers requiring reduction in immunosuppressive dose
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 7

17. Secondary Outcome: BK Nephropathy
Description: The number of patients with BK nephropathy as defined by biopsy. Note that biopsies were not required as part of the study but were only done as part of the patient's standard of care if rejection was suspected (i.e. if the serum creatinine increased by 25% and was not associated with elevated tacrolimus levels or clinical signs of dehydration/illness to account for elevated creatinine)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 0

18. Secondary Outcome: Malignancies
Description: The number of patients developing malignancies including post-transplant lymphoproliferative disorders
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 2

19. Secondary Outcome: Cardiovascular Complications
Description: The number of patients with cardiovascular complications as indicated by conditions such as dysrhythmias, coronary artery disease requiring intervention or myocardial infarction
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 1

20. Secondary Outcome: Development of Donor Specific Antibody
Description: The number of patients with incidence of development of donor specific antibody
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
Number analyzed (Participants) | 50
Participants | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm 1 Everolimus/Reduced Dose Tacrolimus
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 18/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Everolimus/Reduced Dose Tacrolimus (N=50)
Venous thrombosis (Vascular disorders) | 4 (4) — Lower extremity deep venous thrombosis
Pyrexia (General disorders) | 4 (5) — Fever
Influenza A (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2)
Endocarditis (Infections and infestations) | 1 (1) — Aortic endocarditis
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) — UTI - Organism: Escherichia coli
Urinary tract infection (Infections and infestations) | 1 (1) — Escherichia coli UTI
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Increased serum creatinine
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Shortness of breath
Depression suicidal (Psychiatric disorders) | 1 (1) — Depression - suicidal ideation
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — Left arm arteriovenous fistula pseudoaneurysm
Kidney transplant rejection (Immune system disorders) | 1 (1) — Donor specific antibody development (kidney rejection)
Nasal abscess (Infections and infestations) | 1 (1) — Left nostril abscess with facial cellulitis
Parathyroid gland excision (Surgical and medical procedures) | 1 (1) — Subtotal parathyroidectomy classified as serious adverse event due to hospitalization over 24 hours
Nephrectomy (Surgical and medical procedures) | 2 (2) — Bilateral native nephrectomy classified as serious adverse event due to hospitalization over 24 hours
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Everolimus/Reduced Dose Tacrolimus (N=50)
Upper respiratory tract infection (Infections and infestations) | 31 (52)
Urinary tract infection (Infections and infestations) | 9 (19)
Fungal skin infection (Skin and subcutaneous tissue disorders) | 4 (5)
Hyperlipidemia (Metabolism and nutrition disorders) | 14 (14)
Worsening hyperlipidemia (Metabolism and nutrition disorders) | 18 (20)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 18 (25)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Abdominal distention (Gastrointestinal disorders) | 3 (3)
Stomach upset (Gastrointestinal disorders) | 7 (7)
Gastroenteritis (Gastrointestinal disorders) | 3 (3)
Weight gain (Investigations) | 25 (33) — > 10 lbs
Weight loss (Investigations) | 11 (12) — > 10 lbs
Herpes zoster (Infections and infestations) | 5 (5)
Hepatic enzyme increased (Hepatobiliary disorders) | 13 (14)
Stomatitis (Gastrointestinal disorders) | 14 (18) — aphthous mouth ulcers
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3)
Worsening diabetes mellitus (Metabolism and nutrition disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Cellulitis (Infections and infestations) | 3 (3)
Rash, acneiform (Skin and subcutaneous tissue disorders) | 7 (8)
Worsening rash, acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Rash, generalized (Skin and subcutaneous tissue disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Worsening depression (Psychiatric disorders) | 2 (2)
Edema, limb (General disorders) | 23 (30)
Fatigue (General disorders) | 12 (14)
Worsening fatigue (General disorders) | 3 (3)
Blood creatinine increased (Renal and urinary disorders) | 8 (9)
Erythrocytosis (Blood and lymphatic system disorders) | 8 (8) — Post-transplant erythrocytosis
Pyrexia (General disorders) | 9 (9)
Dizziness (Nervous system disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Mental concentration difficulty (Psychiatric disorders) | 3 (3) — Impairment or fogginess
Proteinuria (Renal and urinary disorders) | 11 (12)
Worsening proteinuria (Renal and urinary disorders) | 7 (8)
Chills (General disorders) | 7 (9)
Visual acuity reduced (Eye disorders) | 4 (4)
Generalized body aches (General disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 9 (12)
Worsening leukopenia (Blood and lymphatic system disorders) | 2 (3)
Hyponatremia (Renal and urinary disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Low back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Excessive thirst (Metabolism and nutrition disorders) | 3 (5)
Hematuria (Renal and urinary disorders) | 7 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
BK viremia (Investigations) | 3 (3) — > 500 copies post-transplant
Donor specific antibody positive (Immune system disorders) | 2 (2) — post-transplant
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hypertension (Vascular disorders) | 10 (13)
Worsening hypertension (Vascular disorders) | 9 (9)
Headache (Nervous system disorders) | 8 (11)
Worsening headache (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Worsening dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study is limited by early discontinuation of the 2nd arm in this parallel group study due to safety concerns. All 5 patients with tacrolimus elimination developed donor specific antibodies against DQ-beta HLA antigens and were excluded from study analysis. Protocol section notes enrollment of 55 patients. Results for only 50 patients Due to small sample size, study is not powered to achieve statistical significance.

Statistical significance also impaired without the 2nd arm of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT01935128/Prot_SAP_000.pdf